CLINICAL TRIAL: NCT00585052
Title: A Phase II Study of the Synergistic Interaction of Lovastatin and Paclitaxel For Patients With Refractory or Relapsed Ovarian Cancer
Brief Title: A Phase II Study of Interaction of Lovastatin and Paclitaxel For Patients With Refractory or Relapsed Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, PI left the institution
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Raymond J Hohl, Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200305074
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Epithelial Ovarian Cancer; Lovastatin; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel and lovastatin (Experimental): Paclitaxel given at 80 mg/m2 IV over 1 hour on day 1 and repeated weekly. Lovastatin self-administered at 80mg daily.
  Interventions: Drug: Paclitaxel; Drug: Lovastatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel will be given at 80 mg/m2 IV over 1 hour on day 1 and repeated weekly
  Other Names: Abraxane; Taxol
Drug: Lovastatin — Lovastatin, 80 mg, po, daily will be self-administered by the subject.
  Other Names: Mevacor; Altoprev

SUMMARY:
The purpose of this study is to find out if the treatment combination of paclitaxel and lovastatin is more effective than the currently available chemotherapy for refractory or relapsed ovarian cancer. This research is being done to improve on currently available chemotherapy for ovarian cancer.

DETAILED DESCRIPTION:
The main goal of the study is to find out if adding lovastatin to paclitaxel increases the number of people whose tumors shrink or whose disease responds to the treatment. Another purpose of the study is to find out how long tumors stay reduced in size before growing again as well as how long people live after receiving paclitaxel and lovastatin. The study will also gather information on the side effects, if any, of this combination of paclitaxel and lovastatin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with platinum refractory epithelial ovarian cancer: Defined as those patients with histologically confirmed epithelial ovarian cancer that have not responded (progressive or stable disease as a best response) to an initial chemotherapy regimen that included a platinum agent (cisplatin or carboplatin).
* Patients with platinum resistant ovarian cancer: Defined as those patients with histologically confirmed epithelial ovarian cancer that have relapsed less than 6 months after completion of prior platinum based chemotherapy. If the patient had responded but progressed more than 6 months after completing therapy, the patient must have received at least one additional course of platinum containing chemotherapy or recurred within 6 months of discontinuation of the second-line treatment program.
* Measurable Disease: Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded ) as >/= 20 mm with conventional techniques. The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow up. Image based evaluation is preferred to evaluation by clinical examination. Lesions that are considered to be unmeasurable include the following: bone lesions, leptomeningeal disease, ascites and pleural/pericardial disease.
* Prior treatment with any number of chemotherapeutic regimens is permitted as long as there was an interval of at least 4 weeks since the last chemotherapy.
* Prior treatment with paclitaxel chemotherapy is permitted as long as it was administered on a >/= 3 week regimen and it has been at least 4 weeks since the last treatment.
* Normal Hepatic function
* Total Bilirubin < 2 times upper limits of normal range.
* Transaminases < 2 times upper limits of normal range
* Non-pregnant and non-nursing. Treatment under this protocol would expose an unborn child to significant risks. Women of reproductive potential should agree to use an effective means of birth control.

Exclusion Criteria:

* Other serious illnesses, which would limit survival to <2 years, or a psychiatric condition, which would prevent compliance with treatment or informed consent.
* Performance Status >2
* Uncontrolled or severe cardiovascular disease, diabetes, pulmonary disease, or infection, which in the opinion of the treating physician would make this protocol treatment unreasonably hazardous for the patient.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse within one year.
* Patients who have received any investigational agent within the prior 4 weeks.
* Age < 18 as there is no safety data for lovastatin in this age range.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-08; Primary Completion 2010-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hohl, MD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paclitaxel and Lovastatin
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel and Lovastatin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 61.6 [51 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate of the Combination of Lovastatin and Paclitaxel.
Description: Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >/= 20 mm with conventional techniques. The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow up. Image based evaluation is preferred to evaluation by clinical examination
  * Clinical Examination: Clinically detected lesions will only be considered measurable when they are superficial (e.g. skin nodules and palpable lymph nodes.)
  * Image based evaluation (CT and MRI): Conventional CT and MRI are currently the most reproducible methods of measuring lesions for response assessment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel and Lovastatin
Number analyzed (Participants) | 10
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 0
  Progressive Disease (PD) | 10

2. Secondary Outcome: Time to Progression Using the Combination of Lovastatin and Paclitaxel.
Description: To determine the time to progression using the combination of lovastatin and paclitaxel.
Time Frame: Up to one year
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Paclitaxel and Lovastatin
Number analyzed (Participants) | 10
years | 0.41 (0.202)

ADVERSE EVENTS:
Arm/Group | Paclitaxel and Lovastatin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and Lovastatin (N=10)
Partial small bowel obstruction (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (3)
Increased liver functions (Hepatobiliary disorders) | 1 (1)
Abdominal distention and discomfort (Gastrointestinal disorders) | 1 (1)
Myelodysplasia (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and Lovastatin (N=10)
Nail changes (General disorders) | 3 (3)
Neuropathy (Nervous system disorders) | 7 (16)
Loss of balance (General disorders) | 1 (1)
Sleeplessness (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (6)
Cold (Infections and infestations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sinus infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (16)
Pedal edema (Blood and lymphatic system disorders) | 4 (4)
Eye tearing (Eye disorders) | 2 (2)
Fatigue (General disorders) | 8 (10)
Nausea (Gastrointestinal disorders) | 6 (17)
Headache (General disorders) | 5 (7)
Right upper quadrant pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Alopecia (General disorders) | 9 (10)
Lightheadedness (General disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 8 (8)
Decreased appetite (Gastrointestinal disorders) | 2 (2)
Small bowel obstruction (Gastrointestinal disorders) | 2 (4)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Axillary, benign mass (Blood and lymphatic system disorders) | 1 (1)
Breast, benign mass (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (14)
Side pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 5 (5)
Abdominal cramping/pain (Gastrointestinal disorders) | 7 (15)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 4 (4)
Night sweats (General disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain (General disorders) | 4 (7)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Facial swelling (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Eye/cheek swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal tightness (Gastrointestinal disorders) | 2 (2)
Early satiety/fullness (Gastrointestinal disorders) | 1 (1)
Nail bed fungal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Fingernail/nail bed discoloration (Skin and subcutaneous tissue disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 3 (3)
Burn to fingers (Skin and subcutaneous tissue disorders) | 3 (3)
Leg jumpiness (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Anorexia (Psychiatric disorders) | 1 (2)
Taste disturbance (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Sore tongue (Gastrointestinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Mouth dryness (General disorders) | 1 (1)
Urosepsis (Renal and urinary disorders) | 1 (1)
Lukopenia (Metabolism and nutrition disorders) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder infection (Renal and urinary disorders) | 1 (1)
Itchiness, mild skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Fingernail pain (Skin and subcutaneous tissue disorders) | 1 (1)
Toe pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Ankle edema (Blood and lymphatic system disorders) | 1 (1)
Food allergy (General disorders) | 1 (1)
Bloody nasal drainage (Blood and lymphatic system disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Overheating (General disorders) | 1 (1)
Rhinitis (Infections and infestations) | 2 (3)
Dehydration (General disorders) | 2 (4)
Periorbital edema (Blood and lymphatic system disorders) | 1 (1)
Erythema eyelid (Blood and lymphatic system disorders) | 1 (1)
Nasal drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased oral intake (Gastrointestinal disorders) | 1 (4)
Chills/sweats (General disorders) | 1 (2)
Ankle swelling (Blood and lymphatic system disorders) | 1 (1)
Hand swelling (Blood and lymphatic system disorders) | 1 (1)
Ecchymosis (Blood and lymphatic system disorders) | 1 (1)
Edema (generalized) (Blood and lymphatic system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral edema (Blood and lymphatic system disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (2)
Eyelid irritation (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial closed early due to slow accrual, PI left the institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes